CLINICAL TRIAL: NCT04009720
Title: Repositionable Lotus Edge™ Valve System - Post Market Evaluation of Real World Clinical Outcomes
Brief Title: RESPOND EDGE Post Market Study
Acronym: RESPOND EDGE
Status: Terminated | Type: Observational
Why Stopped: study device Lotus Edge was removed from the market
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2361
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Lotus Edge Device — The LOTUS Edge Valve System is indicated to improve aortic valve function for symptomatic subjects with severe calcific aortic stenosis (aortic valve area [AVA] <1.0 cm2 or AVA index <0.6 cm2/m2) who are at high risk for standard surgical valve replacement.

SUMMARY:
The purpose of the RESPOND EDGE post market study is to collect real world clinical and device performance outcomes data with the Lotus Edge™ Valve System used in routine clinical practice to demonstrate that the commercially available Lotus Edge Valve System is a safe and effective treatment for patients with severe calcific aortic stenosis.

DETAILED DESCRIPTION:
The RESPOND EDGE study is a prospective, open label, single arm, multi-center, observational post market study designed to collect real world clinical and device performance outcomes data of the commercially available Lotus Edge Valve used in routine clinical practice for the treatment of severe calcific aortic stenosis. Approximately 200 real-world, consecutive subjects will be enrolled at up to 20 study centers. The study duration for each subject is expected to be approximately 2 years. Implanted subjects will be contacted for follow-up at 30 days, 1 and 2 years post index procedure. Subjects who are enrolled but not implanted with a Lotus Edge valve will be followed for safety through 30 days after the initial attempted index procedure.

Collection of safety events will include any serious adverse event (SAE), serious adverse device effect (SADE), adverse device effect (ADE), unanticipated serious adverse device effect (USADE), and all Valve Academic Research Consortium (VARC) events regardless of seriousness and device relationship through 2 year follow-up.

ELIGIBILITY:
Subjects will be evaluated for eligibility by the clinical center's heart team per the local standard of practice in accordance with the Directions for Use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who are candidates for Transcatheter Aortic Valve Implantation (TAVI), signed the Informed Consent Form and are selected to receive a LOTUS Edge valve will be evaluated for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
All-cause mortality (Primary Safety Endpoint) | 30 days
  The primary safety endpoint is all-cause mortality at 30 days after the implant procedure. The primary safety endpoint will be evaluated on an intention to- treat (ITT) basis (all subjects enrolled, whether or not a Lotus Edge Valve is implanted).
Mean aortic valve pressure gradient (Primary Effectiveness Endpoint) | Within 7 days after the index procedure (Pre-discharge)
  The primary effectiveness endpoint is the mean aortic valve pressure gradient (mmHg) at pre-discharge as determined by an independent core laboratory. The primary analysis set for the primary effectiveness endpoint is the implanted analysis set.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Dumonteil, MD, Principal Investigator — Clinique Pasteur; Rajesh K Kharbanda, MD, PhD, Principal Investigator — Oxford Heart Centre, John Radcliffe Hospital
Locations (13):
- Rigshospitalet, Copenhagen, Denmark
- University Helsinki, Helsinki, Finland
- Clinique Pasteur, Toulouse, France
- Herzzentrum Universität Leipzig, Leipzig, Germany
- Galway University Hospital, Galway, Ireland
- Az Osp Univ Pisana, Pisa, Italy
- Erasmus MC - Thorax Center, Rotterdam, Netherlands
- University of Lund, Lund, Sweden
- United Kingdom (5):
  - Royal Victoria Belfast, Belfast
  - Royal Sussex County Hospital, Brighton
  - The General Infirmary, Leeds
  - Oxford John Radcliffe Hospital, Oxford
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No